CLINICAL TRIAL: NCT01427946
Title: A Phase 1b/2 Study of Retaspimycin HCl (IPI-504) in Combination With Everolimus in Patients With KRAS Mutant NSCLC
Brief Title: Phase 1b/2 Study of Retaspimycin HCl (IPI-504) in Combination With Everolimus in KRAS Mutant Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-15
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: KRAS mutant; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tanespimycin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retaspimycin HCl (IPI-504) and Everolimus (Experimental): Retaspimycin HCl (IPI-504) and everolimus will be administered on a 21-day cycle. All patients will remain on study until progression of disease or intolerability to study treatments occurs.
  Interventions: Drug: IPI-504; Drug: Everolimus

INTERVENTIONS:
Drug: IPI-504
  Other Names: retaspimycin hydrochloride
Drug: Everolimus
  Other Names: Afinitor

SUMMARY:
Study IPI-504-15 is a Phase 1b/2 clinical trial to evaluate the safety and efficacy of retaspimycin HCl (IPI-504) plus everolimus in patients with KRAS mutant Non-small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase Ib/2 study of retaspimycin HCl (IPI-504) in combination with everolimus. The Phase 1b portion is to test the safety and tolerability of retaspimycin HCl (IPI-504) in combination with everolimus and determine the highest dose of retaspimycin HCl (IPI-504) and everolimus that can safely be given in combination. The Phase 2 portion of this study will continue the evaluation of safety of retaspimycin HCl (IPI-504) in combination with everolimus and compare the effect of the study drugs on tumor response and life expectancy in patients with KRAS mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Voluntarily sign an informed consent form (ICF).
3. Pathological diagnosis of KRAS mutation positive NSCLC - Stage IIIB or IV
4. Archival NSCLC tissue available to provide for analysis or have a lesion that is accessible for biopsy
5. Experienced disease progression during or after receiving at least 1 prior platinum-containing chemotherapy regimen.
6. ECOG performance of 0-1.

Exclusion Criteria:

1. Prior treatment with IPI-504 or other Hsp90 inhibitors.
2. Prior treatment with everolimus, other rapamycin analogs, AP23573(Ridaforolimus), rapamycin, or other mTOR inhibitors.
3. Has not recovered from any toxicities related to prior treatment (to Grade 1 or baseline), excluding alopecia.
4. Inadequate hematologic function defined as:
5. Inadequate hepatic function defined by:
6. Inadequate renal function defined by serum creatinine >1.5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to three years from last patient study visit
  Overall response rate (ORR), defined as a partial response (PR) or complete response (CR) occurring at any point post-treatment according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
Progression Free Survival | Up to three years from last patient study visit
  Progression free survival (PFS), defined as time from study entry to progression or death whichever occurs first.
Time to Progression | Up to three years from last patient study visit
  Time to progression (TTP), defined as time from study entry to progression.
Overall Survival | Up to three years from last patient study visit
  Overall survival (OS), defined as time from study entry to death due to any cause, in patients with KRAS mutant NSCLC administered IPI-504 plus everolimus.

CONTACTS AND LOCATIONS:
Overall Officials: Tess Schmalbach, MD, PhD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - University of Colorado Denver, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York